CLINICAL TRIAL: NCT05468346
Title: Clinical Trial of Absorption, Metabolism and Excretion of [14C]-HEC585 in Chinese Adult Male Healthy Subjects
Brief Title: Study on the Body Mass Balance and Biotransformation of [14C]-HEC585
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEC585-IPF-103
Record Dates: First submitted 2022-05-12; First posted 2022-07-21 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-HEC585 (Experimental): [14C]-HEC585,solid powder，200 mg/100 µCi,single dose，oral
  Interventions: Drug: [14C]-HEC585

INTERVENTIONS:
Drug: [14C]-HEC585 — Single Dose = Solution containing 200 mg/100 µCi [14C]-HEC585

SUMMARY:
This is a single-centre, open-label, non-randomised, single-dose study in healthy male subjects designed to assess the mass balance and biotransformation of [14C]-HEC-585.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males, age: 18 to 45 years old (including the critical value);
2. The body weight is not less than 50 kg, and the body mass index (BMI) is in the range of 19.0~26.0 kg/m2 (including the critical value);
3. Voluntarily participate in this trial, sign the informed consent form before the trial begins, and fully understand the trial content, process and possible risks;
4. Subjects were able to communicate well with investigators and were able to complete the trial as specified in the protocol.

Exclusion Criteria:

1. Comprehensive physical examination, vital signs, laboratory tests [blood routine, blood biochemistry, urine routine, coagulation function, fecal occult blood, thyroid function test (FT3, FT4, TSH)], 12-lead electrocardiogram, X-chest X-ray (frontal) or chest CT, abdominal B-ultrasound (liver, gallbladder, pancreas, spleen and kidneys), new crown screening (nucleic acid + C-reactive protein) and other abnormal and clinically significant examinations;
2. Those who are positive for any one of hepatitis B surface antigen or E antigen, hepatitis C antibody, HIV antibody and syphilis antibody;
3. Those who have taken any drugs that inhibit or induce liver metabolism of drugs within 28 days before screening (see Appendix 1 for details);
4. Use of any prescription or over-the-counter medicines, any vitamin products, health medicines or Chinese herbal medicines within 14 days prior to screening;
5. Those who participated in any clinical trial and received intervention of experimental drugs or medical devices within 3 months before the screening period;
6. Those who have been vaccinated within 1 month before screening or have a vaccination plan during the trial;
7. Have any clinical history of serious diseases or diseases or conditions that the researchers believe may affect the results of the test, including but not limited to the circulatory system, endocrine system, nervous system, digestive system, urinary system or blood, immune, mental and metabolic diseases history;
8. Those who have had heart failure, angina pectoris, myocardial infarction, clinically significant arrhythmia and other heart diseases in the past;
9. Those who have undergone major surgery within 6 months before the screening period or the surgical incision is not completely healed. Major surgery includes but is not limited to any surgery with significant bleeding risk, prolonged general anesthesia, or incision biopsy or obvious traumatic injury ;
10. Abdominal fistula, gastrointestinal perforation or abdominal abscess occurred within 6 months before screening;
11. Have clinically significant bleeding symptoms or a clear bleeding tendency within 3 months before screening, such as gastrointestinal bleeding, hemorrhagic gastric ulcer;
12. Hemorrhoids or perianal diseases with regular/hematochezia, abnormal gastrointestinal function such as irritable bowel syndrome and inflammatory bowel disease, which may affect drug absorption as judged by the researchers;
13. People with allergies, including drug allergies or food allergies, or those who have special requirements for diet and cannot follow a unified diet;
14. Habitual constipation or diarrhea;
15. Binge drinking or frequent drinking within 6 months prior to the screening period, i.e. drinking more than 14 units of alcohol per week (1 unit = 285 mL of beer or 25 mL of 40% alcohol or 100 mL of wine) or alcohol during the screening period Breath test results ≥ 20 mg/dL;
16. Those who smoked more than 5 cigarettes or habitually used nicotine-containing products in the first 3 months of the screening period, and were unable to quit during the trial;
17. Drug abuse or use of soft drugs (such as marijuana) 3 months before the screening period or hard drugs (such as: cocaine, amphetamines, phencyclidine, etc.) 1 year before the screening period, or urine drugs during the screening period ( Drugs) screening test positive;
18. Habitual drinking of grapefruit juice or excessive tea, coffee and/or caffeinated beverages and unable to quit during the trial period;
19. Those with a history of fainting of needles or blood, difficult to collect blood or unable to tolerate venipuncture for blood collection;
20. Workers who need to be exposed to radioactive conditions for a long time, or have significant radioactive exposure (≥2 chest/abdominal CT, or ≥3 other types of X-ray examinations) within 1 year before the test, or have participated in radiopharmaceutical labeling experimenter;
21. Those who have fertility plans during the trial and within 12 months after the administration of the trial drug, or who do not agree that the subjects and their spouses should take strict contraceptive measures during the trial and within 12 months after the administration of the trial drug (see details for details). Appendix 2);
22. Those who have lost blood or donated blood up to 400 mL within 3 months before the screening period, or who have received blood transfusion, or who plan to donate blood within 3 months after the end of this trial;
23. According to the judgment of the investigator, the subject has other factors that make it inappropriate to participate in this trial.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2022-08-14 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
Mass balance | plasma up to 312 hours post dose, urine and fecal samples up to 504 hours post dose
  To determine the mass balance recovery of orally administered [14C]-HEC585

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of HEC-585 and its major metabolites | 312 hours
  Analyze the Peak Plasma Concentration (Cmax) of HEC-585 and its major metabolites (if applicable) to obtain the corresponding pharmacokinetic parameters;
Area under the plasma concentration versus time curve (AUC) of HEC-585 and its major metabolites | 312 hours
  Analyze the Area under the plasma concentration versus time curve (AUC) of HEC-585 and its major metabolites (if applicable) to obtain the corresponding pharmacokinetic parameters;
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 504 hours
  To investigate the safety and tolerability of HEC585 by assessment of Incidence of Treatment-Emergent Adverse Events following administration of of oral dose of 200 mg/100 µCi[14C]-HEC-585

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hutchinson J, Fogarty A, Hubbard R, McKeever T. Global incidence and mortality of idiopathic pulmonary fibrosis: a systematic review. Eur Respir J. 2015 Sep;46(3):795-806. doi: 10.1183/09031936.00185114. Epub 2015 May 14. PMID 25976683
- [Background] Olson AL, Gifford AH, Inase N, Fernandez Perez ER, Suda T. The epidemiology of idiopathic pulmonary fibrosis and interstitial lung diseases at risk of a progressive-fibrosing phenotype. Eur Respir Rev. 2018 Dec 21;27(150):180077. doi: 10.1183/16000617.0077-2018. Print 2018 Dec 31. PMID 30578336
- [Background] Richeldi L, Rubin AS, Avdeev S, Udwadia ZF, Xu ZJ. Idiopathic pulmonary fibrosis in BRIC countries: the cases of Brazil, Russia, India, and China. BMC Med. 2015 Sep 24;13:237. doi: 10.1186/s12916-015-0495-0. PMID 26399999
- [Background] Ingegnoli F, Ughi N, Mihai C. Update on the epidemiology, risk factors, and disease outcomes of systemic sclerosis. Best Pract Res Clin Rheumatol. 2018 Apr;32(2):223-240. doi: 10.1016/j.berh.2018.08.005. Epub 2018 Sep 14. PMID 30527428
- [Background] Hoffmann M, Kasserra C, Reyes J, Schafer P, Kosek J, Capone L, Parton A, Kim-Kang H, Surapaneni S, Kumar G. Absorption, metabolism and excretion of [14C]pomalidomide in humans following oral administration. Cancer Chemother Pharmacol. 2013 Feb;71(2):489-501. doi: 10.1007/s00280-012-2040-6. Epub 2012 Dec 1. PMID 23203815
- [Background] Hoffmann M, Kumar G, Schafer P, Cedzik D, Capone L, Fong KL, Gu Z, Heller D, Feng H, Surapaneni S, Laskin O, Wu A. Disposition, metabolism and mass balance of [(14)C]apremilast following oral administration. Xenobiotica. 2011 Dec;41(12):1063-75. doi: 10.3109/00498254.2011.604745. Epub 2011 Aug 23. PMID 21859393
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30578336/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/26399999/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30527428/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/23203815/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/21859393/